CLINICAL TRIAL: NCT03853460
Title: Bilateral Quadraus LUMBORUM Block in Patients Under Going Cystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, lecturer of anaesthesia and pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: QLMD
Record Dates: First submitted 2019-02-20; First posted 2019-02-25 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: both patients and data collector will be unaware of the group nature
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- epidural group (Active Comparator): ULTRASOUND GUIDED thoracic epidural at T 12 WILL BE INSERTED before anaesthesia induction
  Interventions: Procedure: epidural catheter
- quadus lumborum group (Active Comparator): bilateral ultrasound guided quadratus lumborum catheter will be inserted before anaesthesia induction
  Interventions: Procedure: nerve block catheter

INTERVENTIONS:
Procedure: epidural catheter — ultrasound low frequency probe will be used to determine the depth of the posterior complex to assists placement of midline thoracic epidural
  Arms: epidural group
Procedure: nerve block catheter — ultrasound guided placement of bilateral quadratus lumborum catheters
  Arms: quadus lumborum group

SUMMARY:
ultrasound guided quadratus lumborum will be given for patients under going partial or complete urinary bladder removal.

DETAILED DESCRIPTION:
ultrasound guided quadratus lumborum will be given for patients under going partial or complete urinary bladder removal.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery
* patients between 30 and 60 years

Exclusion Criteria:

* coagulopathy
* infection at insertion site
* patient refusal

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
pain score | 24 hours
  Visual analogue score from 0 to 10 will be used to assess pain postoperative. 0 means no pain. 10 is worst pain

SECONDARY OUTCOMES:
anaesthetic consumption | 4 hours
  calculating the total anaesthetic MAC consumed
diaphragmatic excursion | 24 hours
  assessment of diaphragmatic excursion preoperative and postoperative using low frequency ultrasound probe

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Assiut university, Asyut
  - Faculty of Medicine, Asyut

IPD SHARING:
Plan to Share IPD: No